CLINICAL TRIAL: NCT03778762
Title: Blind Tracheal Intubation Through the Air-Q Intubating Laryngeal Airway in Pediatric Patients. Re-evaluation. A Randomized Controlled Trial.
Brief Title: Re-evaluation of Blind Intubation Through the Air-Q Intubating Laryngeal Airway
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: R/17.11.129
Record Dates: First submitted 2018-12-16; First posted 2018-12-19 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Techniques of Endotracheal Intubation in Pediatrics
Keywords: air-Q, blind intubation, correction maneuvers, fiberoptic guided intubation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blind tracheal intubation through AirQ (Active Comparator): Patients were intubated through the air-Q blindly
  Interventions: Procedure: Blind tracheal intubation through AirQ
- Fiberscopic tracheal intubation through AirQ (Placebo Comparator): Patients were intubated through the air-Q using fibreoptic bronchoscope
  Interventions: Procedure: Fiberscopic tracheal intubation through AirQ

INTERVENTIONS:
Procedure: Blind tracheal intubation through AirQ — underwent blind intubation with correction manoeuvres
  Arms: Blind tracheal intubation through AirQ
Procedure: Fiberscopic tracheal intubation through AirQ — : underwent fibreoptic guided intubation
  Arms: Fiberscopic tracheal intubation through AirQ

SUMMARY:
To compare the success rate of blind technique with correction manoeuvres versus fiber optic- guided Intubation through the air Q laryngeal airway in pediatric patients

DETAILED DESCRIPTION:
A prior G-power analysis was done to estimate the sample size. The primary outcome of this study was the first trial success rate. Using fibre exact test and assuming alpha (type I error) = 0.05 and beta (type II error) = 0.2 (power =80%), 58 patients per group would be sufficient to detect a difference 10 % in success rate among the groups. A drop out 10% of cases was expected; therefore 63 patients were required in each group to detect the difference.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status I-II
* Body weight from 4 to 30 kg

Exclusion Criteria:

* Obesity
* History of gastroesophageal reflux
* History of hyperactive airway
* Patients with congenital disorders associated with difficult airway

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 126 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
The first trial success rate | during first trial of intubation procedure
  percentage of cases of successful tracheal intubation during the first trial

SECONDARY OUTCOMES:
The total success rate | from beginning of manipulation of the endotracheal tube till end of second trial either by successful intubation or failed intubation procedure
  percentage of cases underwent successful tracheal intubation during either first or second trial
Time to ventilation | procedure (Time from beginning of air-Q insertion till full capno-graphic wave)
  time needed to get full capno-graphic waves through connection of air Q to breathing circuit
Time to intubation | procedure (Time from beginning of manipulation of the ETT till full capno-graphic wave)
  time needed to get full capno-graphic waves through connection of endotracheal tube to breathing circuit
Heart rate | After induction of anesthesia till 10 minutes after intubation
Mean arterial blood pressure | After induction of anesthesia till 10 minutes after intubation
blood staining of the device | from extubation till 24 hours after extubation
post-intubation croup | from extubation till 24 hours after extubation
hoarsenes | from extubation till 24 hours after extubation
  and its grade if present Grades of hoarseness: 1=non, 2= mild, 3= moderate, 4= severe)

CONTACTS AND LOCATIONS:
Overall Officials: Enas A Abd el Motlb, MD, Study Chair — Associate Professor
Locations (1):
- Enas A Abd el Motlb, Al Mansurah, DK, Egypt

IPD SHARING:
Plan to Share IPD: Undecided